CLINICAL TRIAL: NCT03480607
Title: Comparative Evaluation of Dexamethasone and Dexmedetomidine as Adjuvants for Bupivacaine in Ultrasound Guided Infraorbital Nerve Block in Infants for Cleft Lip Repair
Brief Title: Dexmedetomidine as Adjuvant for Bupivacaine in Ultrasound Guided Infraorbital Nerve Block for Cleft Lip Repair
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: R/17.05.85
Record Dates: First submitted 2018-03-07; First posted 2018-03-29 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Cleft Lip
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Active Comparator): Dexmedetomidine in conjunction with bupivacaine for infra-orbital nerve block
  Interventions: Drug: Dexmedetomidine group
- Dexamethasone group (Active Comparator): Dexamethasone in conjunction with bupivacaine f
  Interventions: Drug: Dexamethasone group

INTERVENTIONS:
Drug: Dexmedetomidine group — 0.75 ml of 0.5% Bupivacaine in conjunction with 0.5 mcg/kg dexmedetomidine
  Arms: Dexmedetomidine group
Drug: Dexamethasone group — 0.75 ml of 0.5% Bupivacaine in conjunction with 0.1 mcg/kg dexamethasone
  Arms: Dexamethasone group

SUMMARY:
To assess the efﬁcacy of dexamethasone versus dexmedetomidine as adjuncts to bupivacaine for infra-orbital nerve block in infants undergoing cleft lip surgery.

DETAILED DESCRIPTION:
Regarding patient registry; A prior G power analysis was done. Using the results obtained from previous studies and assuming an alpha error of 0.05 and beta error 0f 0.2 (power of the study 80 %), a sample size of 20 patients per group was calculated. A drop out 10% of cases is expected, so; 22 cases per group will be required.

Statistical analysis: Data will be analyzed through SPSS (Statistical Package for Social Sciences). Program version 22. Distribution of data will be first tested by Shapiro test. Data will be presented as mean and standard deviation (SD), median and range or numbers and percentages. For normally distributed data, unpaired t test will be used to compare between mean values of both groups. For pain and sedation scores, Mann Whitney U test will be used. Fisher's exact test will be used for comparison of categorical data. The P value ≤ 0.05 will be considered as the level of statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologist (ASA) physical status I or II

Exclusion Criteria:

* known allergy to any of drugs used
* coagulopathy
* any wound or infection related to puncture site
* major illness
* failure to gain consent of parents.

Ages: 1 Month to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-05-10 (Actual)

PRIMARY OUTCOMES:
Postoperative FLACC scale | for 24 hours after surgery
  FLACC scale: 0 : relaxed/ comfortable, 1-3 : mild discomfort, 4-6 : moderate discomfort, 7- 10: sever discomfort/ Pain / both,
Postoperative sedation score | for 4 hours after surgery
  The degree of sedation will be assessed by using a three point sedation scale based on eye opening: - Alert with spontaneous eye opening 0, - Drowsy with eyes only opening in response to speech 1, - Sedated with eyes opening in response to physical stimulation 2,

SECONDARY OUTCOMES:
Heart rate | For 4 hours after induction
  (beat/min)
Systolic blood pressure | For 4 hours after induction
  (mmHg)
Postoperative nausea | for 24 hours after surgery
  As nausea can't be detected in this age group; so we will detect only if vomiting occur or not and number of attacks.
Haematoma formation after surgery | for 24 hours after surgery
  That will be scored as follows; Yes: there is hematoma formation or No: no hematoma formation
Postoperative vomiting | for 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Enas Abd el Motlb, MD, Study Chair — Mansoura University
Locations (1):
- Mansoura University Childeren Hospital, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided